CLINICAL TRIAL: NCT07234357
Title: Sensory Enrichment Using Aromatherapy for Neurobehavioral and Psychological Symptoms in Early Dementia (SENSE)
Brief Title: Sensory Enrichment Using Aromatherapy for Neurobehavioral and Psychological Symptoms in Early Dementia
Acronym: SENSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Temasek Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/0299
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
Keywords: Aromatherapy; Diffusion Aromatherapy; Essential Oils; Mild Cognitive Impairment (MCI); Mild Dementia; Dementia; Caregiver Burden; Caregiver Stress; Elderly Compliance; Caregiver
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Caregiver Burden | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: Only the intervention group will receive the aromatherapy diffusion, while the control group will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental)
  Interventions: Other: No Intervention
- Intervention Group (Experimental)
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: No Intervention — Participants randomised to the control group will only complete the behavioural and caregiver assessments.
  Arms: Control Group
Other: Aromatherapy — Besides being given assessments mentioned in the control group, participants randomised to the intervention group will be provided with a diffuser, the first batch of the AAPE oil blend (patient to choose 1 out of the 2 blends), and detailed instructions on aromatherapy use. They will be instructed to diffuse 1-2 drops of the oil for 30 minutes in the morning and before bedtime (minimally 5 minutes), inhaling and relaxing during these sessions. An Aromatherapy Diary will be provided to track daily compliance, record adverse events, and document the number of minutes used each night.
  Arms: Intervention Group

SUMMARY:
To determine if diffusion aromatherapy exposure to an essential oil blend can potentially improve mild cognitive impairment/mild dementia symptoms and relieve caregiver stress.

This study also allows us to gauge the willingness of elderly patients in complying with long-term aromatherapy treatments.

DETAILED DESCRIPTION:
SENSE is a non-blinded study that aims to recruit 200 participants, consisting of 200 patients with MCI or mild dementia, along with their respective caregivers. Participants will be recruited from the Geriatric Clinic in Sengkang General Hospital, in either English or Chinese. Participants are randomized into the control and intervention group, in which the latter will receive an aromatherapy diffuser, a proprietary aromatic asian plant extract (AAPE) as an essential oil blend to add into the diffuser, and an aromatherapy diary to fill up for 6 months. The participants of the intervention group are to diffuse the essential oils twice daily for a minimum of 5 minutes each session, and will also receive phone calls at the 2, 4, 6, 8, 16, and 20th week timepoint to check on compliance and adverse events.

Both the control and intervention group will complete questionnaires on the first visit, mid-intervention visit (12th week timepoint) and final visit (24th week timepoint):

Patients:

* Patient Baseline Data Collection Form (only for first visit)
* Mini-mental state examination (MMSE)
* Cornell Scale for Depression in Dementia (CSDD)
* Rating Anxiety in Dementia (RAID)
* Sniffin' Sticks Olfactory Test (only for first and final visit)

Caregivers:

* Caregiver Baseline Data Collection Form (CBDCF)
* Neuropsychiatric Inventory Questionnaire (NPI-Q)
* ZBI-12 (Zarit Caregiver Burden Assessment)

All three visits are physical visits at Sengkang General Hospital. Upon completion of each physical visit's requirements, participants will receive a $10 reimbursement voucher.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Aged 50 years old and above.
* Confirmed diagnosis of MCI or mild dementia based on clinical records.
* Has one identified caregiver aged 21 years and above who is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥2 hours/day ≥3 days/week; agrees to accompany the subject to each study visit; and is able to verify daily compliance with study intervention.

For caregivers:

* Aged 21 years old and above.
* Willing and able to provide written informed consent
* Identified as the caregiver for recruited patient in this study can read, understand, and speak the designated language at the study site; either lives with the recruited patients or sees the patient for ≥2 hours/day ≥3 days/week.
* Agrees to accompany the patient to each study visit; and can verify daily compliance with study intervention.

Exclusion Criteria:

For patients:

* Olfactory impaired/dysfunctional.
* Known or suspected hypersensitivity/allergy to essential oils or any components of the formulations.
* Has Reactive Airway Disease (e.g, Asthma).
* Participant without a caregiver.
* Pregnant, breastfeeding, or intending to conceive during study period.

For caregivers:

* Physically or mentally incapable of providing verbal / written consent
* Does not have regular or meaningful contact with the participant (e.g. less than 2 hours/day or less than 3 days/week).
* Not able to follow patient to each study visit.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of an olfactory enrichment program in improving the well-being of patients with mild cognitive impairment (MCI) and dementia. | Mid-intervention (12 weeks), and post intervention (24 weeks).
  To gauge the compliance and willingness to comply with long-term aromatherapy treatments in their homes, in a local context.
  Compliance rate will be calculated using the total number of sessions that the participants have fulfilled, for at least 5 minutes each session.
  Patients that are unable to meet the minimum of 50% compliance will be withdrawn from the study.
Preliminary efficacy of the intervention in reducing Behavioural and Psychological Symptoms of Dementia (BPSD) to inform sample size calculations for a larger study through the use of Rating Anxiety in Dementia (RAID) Questionnaire. | Baseline (first visit), mid-intervention (12 weeks), and post intervention (24 weeks).
  RAID utilizes a scale that includes "unable to evaluate" and 0-3. Questionnaires are analysed by tabulating the total scores of each questionnaire to assess the severity of anxiety.
Preliminary efficacy of the intervention in reducing Behavioural and Psychological Symptoms of Dementia (BPSD) to inform sample size calculations for a larger study through the use of Cornell Scale for Depression in Dementia (CSDD) Questionnaire. | Baseline (first visit), mid-intervention (12 weeks), and post intervention (24 weeks).
  CSDD utilizes a scale that includes "absent" and 0-2. Questionnaires are analysed by tabulating the total scores of each questionnaire to assess the severity of depressive symptoms.

SECONDARY OUTCOMES:
Preliminary efficacy of the intervention in maintaining cognitive function in patients with MCI and dementia. | Baseline (first visit), mid-intervention (12 weeks), and post intervention (24 weeks).
  This is measured using Mini-mental state examination (MMSE), which measures cognitive function on a 30-point scale. A higher score indicates better cognitive function.
Impact of the intervention on caregiver stress and burden via Neuropsychiatric Inventory Questionnaire (NPI-Q) | Baseline (first visit), mid-intervention (12 weeks), and post intervention (24 weeks).
  For the caregivers to fill, to see if the impact of diffusion aromatherapy on the respective patients can improve behavioural symptoms observed in the patient. The NPI-Q requires rating presence of a symptom (a "yes" or "no" screening question), the severity on a 1-3 point scale, and caregiver's distress from the symptom on a 0-5 point scale. The total scores of these questionnaires help to assess the severity of caregiver stress and burden, with a higher total score suggesting overall a greater presence of neuropsychiatric symptoms.
Impact of the intervention on caregiver stress and burden via ZBI-12 (Zarit Caregiver Burden Assessment) | Baseline (first visit), mid-intervention (12 weeks), and post intervention (24 weeks).
  For the caregivers to fill, to see if the impact of diffusion aromatherapy on the respective patients can potentially relieve some caregiver stress and burden. The ZBI-12 is completed by the caregivers and utilises a 0-4 point scoring system for 12 questions totaling a score from 0 to 48, where higher scores indicate greater caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Teh Bin Tean, MBBS, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided